CLINICAL TRIAL: NCT01737892
Title: Assessment and Evaluation of Pharmacokinetic Profile of E004 in Healthy Adults (A Randomized, Evaluator-Blind, Single-Dose, Two Arm, Crossover, PK Study in Healthy Volunteers)
Brief Title: Assessment and Evaluation of Pharmacokinetic Profile of E004 in Healthy Adults
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: unable to validate analytical method
Sponsor: Amphastar Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: API-E004-CL-B4
Record Dates: First submitted 2012-11-20; First posted 2012-11-30 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-02

CONDITIONS: Asthma
Keywords: Asthma; Pharmacokinetics; Epinephrine; Bronchodilator; Metered dose inhaler
MeSH Terms: conditions — Asthma | interventions — Epinephrine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm T-Epinephrine Inhalation Aerosol HFA (Experimental): Experimental arm utilizing Epinephrine HFA-MDI (E004)
  Interventions: Drug: Arm T Epinephrine Inhalation Aerosol HFA, 125 mcg, 1 inhalation
- Arm C-Epinephrine Inhalation Aerosol CFC (Active Comparator): Active comparator arm utilizing Epinephrine CFC-MDI
  Interventions: Drug: Arm C-Epinephrine Inhalation Aerosol CFC

INTERVENTIONS:
Drug: Arm T Epinephrine Inhalation Aerosol HFA, 125 mcg, 1 inhalation — Epinephrine Inhalation Aerosol HFA, Single dose 125 mcg, 1 inhalation
  Arms: Arm T-Epinephrine Inhalation Aerosol HFA
Drug: Arm C-Epinephrine Inhalation Aerosol CFC — Epinephrine Inhalation Aerosol - CFC, Single dose 220 mcg, 1 inhalation
  Other Names: Primatene Mist
  Arms: Arm C-Epinephrine Inhalation Aerosol CFC

SUMMARY:
This study examines the pharmacokinetic profile of Armstrong's proposed Epinephrine Inhalation Aerosol USP, an HFA-MDI (E004), using a stable isotope deuterium-labeled epinephrine (epinephrine-d3) to differentiate the administered drug from the endogenous epinephrine, in healthy male and female adult volunteers. The current study is designed to complement an earlier PK study, API-E004-CL-B, for a more thorough evaluation of the E004 PK. Safety of E004 will also be evaluated.

DETAILED DESCRIPTION:
This study is a randomized, evaluator-blind, single dose, two-arm, crossover, PK study, to be conducted in ~18 healthy, male and female, adult volunteers. PK will be studied using E004-d3 at 125 mcg per inhalation (Arm T). A previously marketed Epinephrine CFC-MDI, labeled "For Investigational Use Only" will be used as a Reference Control (Arm C).

The main features of the study design are:

(1) All candidates must be screened and must satisfy all enrollment criteria. All enrolled subjects will participate in two Study Visits, corresponding to two randomized treatments. Each Study Visit consists of a pre-dose baseline assessment and a post-dose evaluation for 6 hours.

(2) It is important to minimize physical and psychological disturbances to the endogenous epinephrine concentrations in the study subjects, before and during the study visits. All subjects must maintain a reclining or recumbent resting position during the entire Study Visit, with physical activities restricted to a minimum necessity for bathroom trips and study activities. Caffeine-containing (including de-caffeinated) foods or beverages are prohibited. Physical exercise, unnecessary physical activities, and video games are prohibited throughout the study visit.

(3)At the Screening Visit and the beginning of each Study Visit, each subject will be trained on the correct self-administration of MDI, using a simulation MDI unit that contains no active drug. The following two randomized treatments will be self-administered at two Study Visits:

Treatment T: Two (2) inhalations of E004-d3 (125 mcg/inhalation), totaling 250 mcg of epinephrine-d3;

Treatment C: Two (2) inhalations of Epinephrine CFC-MDI (220 mcg/inhalation, totaling 440 mcg of epinephrine base equivalent).

(4) PK blood samples will be taken from a vein in a hand or arm via an indwelling anticoagulated IV catheter, or by venipunctures, at scheduled time points of predose baseline (within 30 minutes of dosing), and at 2±1, 5±1, 7.5±1, 10±1, 12.5, 15, 20, 25, 30, 45, 60, 90, 120, 240 and 360 minutes postdose. The total volume of blood taken per subject shall not exceed 500 mL in any 30-day period. Study visit schedule may be adjusted to avoid overdrawing blood in any 30-day period.

(5) At each PK sampling point, blood samples (~ 5mL), will be collected in ice-chilled potassium-EDTA sample tubes, each containing pre-added 1% (V:V) of a 1.0 M sodium metabisulfite solution as an antioxidant. Sample tubes will be labeled with a sample ID# (consisting of subject ID#, Study Visit#, and sample#). The sample tubes will be kept on ice or refrigerated, and will be centrifuged within 60 minutes of collection. The harvested plasma from each sample tube will be transferred to, and stored in, 2 storage tubes, respectively, and frozen at NMT -20 degrees C until analysis.

(6) PK samples will be analyzed with an established LC/MS/MS method, with a quantitative detection limit of 5 pg/mL, for both epinephrine-d3 (MW=186) and epinephrine (MW=183).

(7) Safety parameters and adverse drug events, if any, will be monitored and documented at each study visit. An End-of-Study (EOS) safety evaluation will be conducted at the end of, or within 7 days after, Study Visit-2.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy, male and female adults, 18-30 yrs of age at Screening
* Having no clinically significant respiratory, cardiovascular and other systemic or organic illnesses, per investigator discretion;
* Body weight greater than or equal to 50 kg for men and greater than or equal to 45 kg for women, and BMI within the range of 18.5 - 30.0 kg/m2 inclusive
* Sitting blood pressure less than or equal to 135/90 mmHg;
* Demonstrating negative alcohol/drug screen tests;
* Demonstrating negative HIV, HBsAg and HCV-Ab screen tests;
* Women of child-bearing potential must be non-pregnant, non-lactating, and practicing a clinically acceptable form of birth control;
* Having properly consented and satisfied all other inclusion/exclusion criteria as required for this protocol.

Exclusion Criteria:

* A smoking history of more than or equal to 10 pack-years, or having smoked within 6 months prior to Screening;
* Upper respiratory tract infections within 2 weeks, or lower respiratory tract infection within 4 weeks, prior to Screening
* Any current or recent respiratory conditions that, per investigator discretion, might significantly affect pharmacodynamic response to the study drugs, including but not limited to: asthma, COPD, cystic fibrosis, bronchiectasis, tuberculosis, emphysema, etc.
* Concurrent clinically significant cardiovascular, hematological, renal, neurologic, hepatic, endocrine (including diabetes), psychiatric, neoplastic or other illnesses that in the opinion of the investigator could impact on the conduct, safety and evaluation of the study
* Known intolerance or hypersensitivity to any of the study MDI ingredients (i.e., epinephrine, HFA-134a, CFC-12, CFC-114, polysorbate-80, ethanol, thymol, nitric acid and ascorbic acid)
* Use of prohibited drugs or failure to observe the drug washout restrictions
* Having been on other investigational drug/device studies, or donated blood, in the last 30 days prior to Screening.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2012-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Calculation and Comparison of relative Bioavailability of Epinephrine | up to 30 min predose and at 2, 5, 7.5, 10, 12.5, 15, 20, 25, 30, 45, 60, 90, 120, 240 and 360 minutes postdose
  Blood PK samples will be collected at each visit for both study arms, then the Area Under the Curve (s) will be calculated for both arms and compared to give relative bioavailability

SECONDARY OUTCOMES:
Vital Signs | up to 30 min predose and at 2, 5, 7.5, 10, 12.5, 15, 20, 25, 30, 45, 60, 90, 120, 240 and 360 minutes postdose
  Vital signs (SBP/DBP, blood pressure and heart rate) will be documented and summarized
12-lead ECG (Routine and QT/QTc analysis) | up to 30 min predose and at 5, 10, 15, 20, 30, 60, 120, and 360 minutes postdose
  A 12-lead ECG (Routine and QT/QTc analysis) will be documented.
Physical Examinations | up to 30 min predose and after 360 min post last dose
  Physical examinations will be documented at screening and end of study
Lab tests | up to 30 min predose
  Lab tests, including CBC, serum comprehensive metabolic panel, urinalysis, and drug/alcohol screens for all subjects and urinary pregnancy test for women of child-bearing potential will be performed and documented

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Evilevitch, M.D., Study Director — Amphastar Pharmaceuticals, Inc.
Locations (1):
- West Coast Clinical Trials, LLC, Cypress, California, United States

REFERENCES:
- [Background] Pinnas JL, Schachtel BP, Chen TM, Roseberry HR, Thoden WR. Inhaled epinephrine and oral theophylline-ephedrine in the treatment of asthma. J Clin Pharmacol. 1991 Mar;31(3):243-7. doi: 10.1002/j.1552-4604.1991.tb04969.x. PMID 2019665
- [Background] Hendeles L, Marshik PL, Ahrens R, Kifle Y, Shuster J. Response to nonprescription epinephrine inhaler during nocturnal asthma. Ann Allergy Asthma Immunol. 2005 Dec;95(6):530-4. doi: 10.1016/S1081-1206(10)61014-9. PMID 16400891
- [Background] Warren JB, Doble N, Dalton N, Ewan PW. Systemic absorption of inhaled epinephrine. Clin Pharmacol Ther. 1986 Dec;40(6):673-8. doi: 10.1038/clpt.1986.243. PMID 3780129
- [Background] Cripps A, Riebe M, Schulze M, Woodhouse R. Pharmaceutical transition to non-CFC pressurized metered dose inhalers. Respir Med. 2000 Jun;94 Suppl B:S3-9. PMID 10919679
- [Background] Dickinson BD, Altman RD, Deitchman SD, Champion HC. Safety of over-the-counter inhalers for asthma: report of the council on scientific affairs. Chest. 2000 Aug;118(2):522-6. doi: 10.1378/chest.118.2.522. PMID 10936150
- [Background] Kushner DJ, Baker A, Dunstall TG. Pharmacological uses and perspectives of heavy water and deuterated compounds. Can J Physiol Pharmacol. 1999 Feb;77(2):79-88. PMID 10535697